CLINICAL TRIAL: NCT01693874
Title: Mindfulness-based Stress Reduction and Cognitive Function in Stress and Aging
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Eric Lenze, Professor of Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AT007064
Record Dates: First submitted 2012-03-29; First posted 2012-09-26 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Anxiety Disorders; Depression
Keywords: anxiety; depression; cognition; MBSR; mindfulness; stress; elderly
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness Based Stress Reduction (Experimental): All participants in this arm receive Mindfulness Based Stress Reduction (MBSR).
  Interventions: Behavioral: MBSR
- control (Active Comparator): All participants in this arm receive an attention control
  Interventions: Behavioral: control (health education)

INTERVENTIONS:
Behavioral: MBSR — Mindfulness-Based Stress Reduction
  Arms: Mindfulness Based Stress Reduction
Behavioral: control (health education) — health education
  Arms: control

SUMMARY:
The investigators are developing and then testing whether Mindfulness-Based Stress Reduction, a group-based instruction for increasing mindfulness, reduces anxiety and depressive symptoms and improves cognitive functioning in older adults.

ELIGIBILITY:
Inclusion Criteria:

* aged 65+
* current depressive and/or anxiety symptoms
* current depressive and/or anxiety disorder
* able to participate in behavioral study

Exclusion Criteria:

* unable to participate in study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 103 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
cognitive functioning | approximately 2 months of study intervention
  neuropsychological battery examining memory, executive functioning, and attention

SECONDARY OUTCOMES:
mind-wandering | 2 months of intervention
  computerized task(s) of mind-wandering
mindfulness | 2 months of intervention
  self-report plus ecological momentary assessment measurements of mindfulness (process variable).
anxiety and depressive symptoms | 2 months of intervention
  scales of self-report anxiety and depressive symptoms from NIH PROMIS, and worry severity (Penn State Worry Questionnaire Abbreviated). also we will examine ecological momentary assessment measurements of anxiety and depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lenze, MD, Principal Investigator — Washington University School of Medicine; Julie Wetherell, PhD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California San Diego, San Diego, California
  - Washington University School of Medicine, St Louis, Missouri

REFERENCES:
- [Derived] Kornfield SL, Nicol GE, Lenze EJ, Yingling M, Loebach Wetherell J. Mindfulness-Based Stress Reduction in Older Individuals: Who Benefits the Most? Adv Mind Body Med. 2022 Winter;36(1):4-12. PMID 35476747
- [Derived] Haddad R, Lenze EJ, Nicol G, Miller JP, Yingling M, Wetherell JL. Does patient expectancy account for the cognitive and clinical benefits of mindfulness training in older adults? Int J Geriatr Psychiatry. 2020 Jun;35(6):626-632. doi: 10.1002/gps.5279. Epub 2020 Mar 20. PMID 32017250
- [Derived] Wetherell JL, Hershey T, Hickman S, Tate SR, Dixon D, Bower ES, Lenze EJ. Mindfulness-Based Stress Reduction for Older Adults With Stress Disorders and Neurocognitive Difficulties: A Randomized Controlled Trial. J Clin Psychiatry. 2017 Jul;78(7):e734-e743. doi: 10.4088/JCP.16m10947. PMID 28686822